CLINICAL TRIAL: NCT05107323
Title: Compassionate Schools: Feasibility and Effectiveness Study of a Compassionate Mind Training Program to Promote Teachers Wellbeing
Brief Title: Feasibility and Effectiveness Study of a Compassionate Mind Training Program for Teachers
Acronym: COMP-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Compassionate Mind Foundation (Unknown); Reed Foundation (Unknown)
Responsible Party: Principal Investigator, Marcela Matos, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CINEICC-01-MM
Record Dates: First submitted 2021-10-19; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Teachers
Keywords: Compassionate Mind Training; Teachers; Feasibility study; Effectiveness study; Psychophysiological wellbeing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMT-T (Experimental): The CMT-T is a Compassionate Mind Training program tailored for teachers, delivered in a group format across eight sessions of approximately 2.5 hours each. In each session, besides presenting relevant theoretical constructs addressed in that session, participants are invited to complete experiential exercises, compassion and mindfulness meditation practices, and work in small groups to share their experiences, followed by a plenary session. There are six different modules addressed during the 8-sessions CMT-T
  Interventions: Behavioral: Compassionate Mind Training for Teachers
- Waiting list (No Intervention): Participants in the waiting list control group were not offered an intervention.

INTERVENTIONS:
Behavioral: Compassionate Mind Training for Teachers — Compassionate Mind Training for Teachers is a biopsychosocial evidence-based approach that aims to foster compassion, affect regulation, prosocial qualities and wellbeing in teachers.
  Arms: CMT-T

SUMMARY:
Given the growing research on the multidimensional benefits of compassion cultivation, the current study sought to explore the feasibility and effectiveness of a Compassionate Mind Training intervention for Teachers (CMT-T) on teachers' psychological distress, wellbeing and compassion to self and others using a randomised controlled and stepped wedge design. The CMT-T specifically aimed at promoting positive affect and satisfaction with professional life and reducing symptoms of depression, anxiety, stress, and burnout, by increasing the flows of compassion (for self, for others and from others), self-compassion and compassion to others motivations and actions, and by diminishing fears of compassion (for self, for others and from others) and self-criticism. Furthermore, the present study aimed to explore the impact of the CMT-T on heart rate variability (HRV), an indicator of vagal regulatory activity and a physiological marker of a person's ability to flexibly respond to environmental challenges and regulate emotional responses. In light of previous research pointing to the role of individual differences in self-criticism on how individuals respond to compassion-based interventions, this study aimed to examine how self-criticism would influence the effects of the CMT-T intervention. Baseline self-criticism was hypothesized to impact the CMT-T effects on the primary and secondary outcome variables. In addition, the current study aimed to examine whether the effects of attending the CMT-T were sustained at 3-month post-intervention. Given that the inter-relationship between the three flows of compassion (i.e., compassion for others, being open to compassion from others, and self-compassion) is a key aspect of the CMT approach, the study sought to explore whether the associations between the flows of compassion would change from before to after the CMT-T, particularly whether these were strengthened after training. Finally, this study aimed to examine the mechanisms of change for the primary outcome variables at post-intervention. It is hypothesized that the changes occurred after the CMT-T intervention were mediated by changes in competencies for compassion for self, for others and from others, decreased levels fears of compassion for self, from others and from others, enhanced affect regulation, diminished self-criticism.

DETAILED DESCRIPTION:
The main aim of COMP-S is to test the impact of a compassionate mind training intervention for teachers: CMT-T on indicators of mental, physiological and professional wellbeing.

The major goals of this project are to:

1. Test the effects of the CMT-T on psychological primary outcomes (i.e. overall positive affect, symptoms of depression, anxiety and stress, burnout and professional wellbeing) and secondary outcomes (i.e. compassion, fears of compassion, self-criticism, affect regulation).
2. Test the impact of the CMT-T on autonomic (i.e. heart-rate variability) biomarkers related to positive affect systems linked to affiliation and prosociality;
3. Test the mediator effect of changes in the psychological processes targeted by the intervention (i.e. secondary outcomes: compassion, fears of compassion, self-criticism, affect regulation) on the impact of the CMT-T on the primary psychological outcomes, and on the biophysiological markers.
4. Investigate the moderator effect of baseline individual differences in self-criticism, depressive symptoms and sociodemographic variables (i.e. age, gender) and occurrence of major life events, on the impact of the CMT-T on the psychological and biophysiological outcomes.
5. Assess the moderator effect of practice frequency and helpfulness, and embodiment of compassionate qualities on everyday life, on the impact of the CMT-T on the psychological and biophysiological outcomes.

STUDY DESIGN The study was a two-arm randomized controlled trial (RCT), with one intervention group (CMT-T) and one waitlist control group (WLC), and a stepped-wedge design where all groups and participants in groups were offered the intervention. Prior to data collection, the study was approved by the Ethics Committee of the Faculty of Psychology and Educational Sciences of the University of Coimbra (CEDI22.03.2018).

Given the stepped wedge design, there were four assessment moments in the study: 1) Time 1 (T1) - baseline/pre-intervention assessment, was completed by the CMT-T group and the WLC group during the week previous to the start of the CMT-T intervention; 2) Time 2 (T2) - post-intervention assessment one was completed by CMT-T group and WLC group during the first-week post-intervention; 3) Time 3 (T3) - post-intervention assessment two, was completed by WLC group participants one week after they had also received the CMT-T intervention; 4) 3-months Follow-up assessment, this was conducted three months after the CMT-T conclusion (for all participants who completed the intervention). In T1, T2, and T3 all participants completed a set of self-report questionnaires. A subsample of participants from both conditions underwent the HRV measurement at T1, T2, and T3. In the 3-month follow-up assessment, only self-report data were collected.

PARTICIPANTS AND RECRUITMENT Participants were eligible for participation if they: (a) were teachers in the enrolled schools; and (b) provided informed consent. Participants were recruited amongst teaching staff in public schools (pre to high school grades) in the centre region of Portugal. Schools' boards were invited to participate in the study. With their authorization, a 2-hour recruitment session was conducted at the school and all teaching staff invited by the board. The session included a brief description of the study aims, procedures and ethical considerations. Teachers interested in participating provided their contact information. They were then contacted via email assessed for inclusion criteria and required to provide informed consent. Informed consent clarified the voluntary, confidential and anonymous nature of the study and data protection rights. Participants who meet the eligibility criteria to enter the study were randomly assigned within each school (using a computer-based random allocation) to either the CMT-T intervention or the waitlist control (WLC) group. The WLC group started the CMT-T after the first CMT-T group had completed the intervention. In total, six groups received the CMT-T, which was delivered in the school setting.

INTERVENTION The Compassionate Mind Training Program for Teachers (CMT-T) is a psychological intervention program delivered in a group format across eight sessions of approximately 2.5 hours each. In each session, besides presenting relevant theoretical constructs addressed in that session, participants are invited to complete experiential exercises, compassion and mindfulness meditation practices, and work in small groups to share their experiences, followed by a plenary session. There are six different modules addressed during the 8-sessions CMT-T.

Teachers attending the 8-week CMT-T were invited to practice the CMT-T exercises daily. In addition to self-report measures, teachers were asked to complete weekly Practice Diaries and Session Evaluation forms. Access to the Project website (https://escolascompassivas.wixsite.com/cmtescolas) allowed participants further information about the program, psychoeducation information and materials, practices instructions and audio files containing the meditation practices. Weekly gentle reminder emails were sent to participants motivating them to practice the exercises. A final CMT and Forest Bathing 1-day retreat was held at the end of the intervention.

DATA ANALYSIS Power analysis was calculated at priori using G*Power 3.1 for Analysis of Variance (ANOVA). Results indicated that a sample size of 27 per group (n = 54) was needed, using a significance level of .05 and a power of 95% to detect significant fixed effects, main effects, and interaction effects, with a large effect size (f = 0.25).

All data analyses were performed using IBM SPSS Statistics for Windows (Version 27.0), and the alpha level was set at .05. For continuous variables, independent samples t-tests were conducted, and for categorical variables, chi-square tests were performed.

To examine mean differences between pre-intervention (T1) and post-intervention (T2) in the primary and secondary outcome variables, a series of 2 (condition) × 2 (time) repeated measures ANOVAs were performed. To examine the mean differences in the study variables within each group, a series of repeated measures ANOVAs were conducted for each group comparing pre and post-intervention. For ANOVAs, effect sizes were calculated using partial eta square (ƞ2p). For independent and paired-samples t-tests, effect sizes were calculated using Cohen's d. A confidence interval of 95% was used in all the analyses. A stepped wedge analysis was performed in the subgroup of participants who participated in the WLC group between T1 and T2 and then completed the CMT-T between T2 and T3. Repeated Measures ANOVAs were performed to test differences in all study's variables from baseline to pre-intervention and post-intervention. Post-Hoc analyses were used to explore pairwise differences (baseline-to-pre-intervention; baseline-to-post-intervention, and pre-to-post-intervention).

To assess whether the post-CMT results were maintained, repeated measures ANOVAs were computed to test for mean differences between post-treatment (T2) and 3-months follow-up (T3). Pearson product-moment correlation analyses were calculated to explore whether the CMT-T would strengthen the associations between the three flows of compassion from pre- to post-intervention in all participants who completed the CMT-T.

Finally, to explore the psychological processes that underlie the changes in the primary outcomes after the CMT-T intervention MEMORE macro (Mediation and Moderation analysis for Repeated measures designs) was used. MEMORE allows for the estimation of total, direct, and indirect effects of independent variable (X) on dependent variable (Y) through one or more mediators (M) simultaneously two-occasion within-subjects design.

ELIGIBILITY:
Inclusion Criteria:

* being a teacher in the enrolled schools
* provide informed consent

Exclusion Criteria:

* not being a teacher in the enrolled schools
* not provide informed consent

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in positive affect | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Types of Positive Affect Scale (TPAS). The TPAS is an 18-item scale that measures the degree to which people experience different positive emotions. Each item is rated on a 5-point scale (ranging from 0 to 4). Higher scores mean higher levels of positive affect.
Changes in satisfaction with teachers' professional life | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Satisfaction with Teachers' Professional Life (SWTPL). The SWTPL is a 5-item scale aimed to assess global satisfaction with teachers' professional life. Each item is rated on a 5 Likert-type scale, ranging from I completely disagree (1) to I completely agree (5). Higher scores reflect higher satisfaction with teachers' life.
Changes in symptoms of depression, anxiety and stress | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Depression, Anxiety and Stress Scales-21(DASS-21). The DASS-21 is a self-report instrument comprising three subscales that address depressive (seven items), anxiety (seven items) and stress symptoms (seven items). Participants are asked to rate the frequency of symptoms during the previous week using a 4-point scale from did not apply to me at all (0) to applied to me very much, or most of the time (3). Higher scores in the each subscale indicate higher levels of depressive, anxiety or stress symptoms.
Changes in burnout | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Shirom-Melamed Burnout Measure (SMBM). The SMBM is a 14-items self-report measure addressing work-related burnout using a 7-point scale, ranging from never (1) to always (7). The SMBM comprises three dimensions associated with work: physical exhaustion, cognitive weariness, and emotional exhaustion, with higher scores reflecting greater burnout symptoms.

SECONDARY OUTCOMES:
Changes in the flows of compassion (self-compassion, compassion to others and compassion from others) | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Compassionate Engagement and Action Scales (CEAS). The CEAS assesses the three flows of compassion according to Gilbert's evolutionary multidimensional model of compassion and the Compassion Focused Therapy framework: 1) Self-compassion, 2) Compassion for others, 3) Compassion from others. Items are rated according to the frequency of responding to one's own suffering, others' suffering or the experience of receiving compassion from others. A response scale ranging from never (1) to always (10) is used for rating the items. Higher scores e each scale reflect higher compassion for self, for others and from others (respectively).
Changes in self-compassion and compassion to others motivation and action | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Compassion Motivation and Action Scales (CMAS) The CMAS is a 30-item self-report measure designed to be specifically used as a measure of the change in compassionate motivation and action over time. The self-compassion dimension encompasses 18 items, the compassion to others dimension includes 12 items. A 7-point scale ranging from completely disagree (1) to completely agree (7) is used to rate each item. Higher scores in each dimension mean elevated levels of self-compassion and compassion to others motivation and action.
Changes in fears of compassion (for self, for others, from others) | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Fears of Compassion Scale (FoC). The FoC is a broadly used self-report measure of fears, blocks and resistances to compassion. It assesses barriers to giving compassion to others (10 items), receiving compassion from others (13 items), and being self-compassionate (15 items). The 38 items are answered on a 5-point Likert scale ranging from don't agree at all (0) to completely agree (4). Higher scores reflect higher fears of compassion (for self, for others, from others).
Changes in self-criticism | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Forms of Self-Criticism and Self-Reassurance Scale (FSCRS). The FSCRS is a 22-items self-report instrument assessing how one thinks and reacts when dealing with failures or setbacks. The FSCRS encompasses two forms of self-criticism: (1) inadequate-self and (2) hated-self and (3) assesses the ability to be self-reassuring. Respondents are asked to choose in a 5-point scale, ranging from not at all like me (0) to extremely like me (4), the degree to which each item relates to their own experience. Higher scores on the self-criticism subscales indicate higher levels of self-criticism.
Changes in perceived emotional climate at work | up to 6 months (from baseline to 3-months follow-up)
  Assessed by the Emotional Climate in Organizations Scales (ECOS). ECOS was developed based on the affect regulation systems model proposed by Gilbert (106) and assesses the presence/activation of the three affect regulation systems: threat, drive, soothing/safeness. Each scale comprises 15 items (five items for each type of emotion system), rated in a 5-point Likert-type scale scored between never (0) and always (4). Higher scores are indicative of higher levels of threat, drive or soothing/safeness emotions at work.

OTHER OUTCOMES:
Changes in Heart-rate variability (HRV) | up to 10 weeks (from baseline to post-intervention)
  For the measurement of HRV, the electrocardiogram (ECG) was recorded using Firstbeat Bodyguard2 (Firstbeat Technologies Ltd.) with a standard electrode configuration (right clavicle and precordial site V6). Heart rate and a time domain measure of HRV (Root Mean Square Successive Difference; RMSSD) were then obtained for pre- and post-intervention in both groups. According to the Task Force guidelines, the RMSSD reflects the integrity of vagus nerve-mediated autonomic control of the heart.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gilbert, PhD, OBE, Study Chair — University of Derby; Compassionate Mind Foundation
Locations (1):
- Center for Research in Neuropsychology and Cognitive and Behavioural Intervention (CINEICC), Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matos, M., Palmeira, L., Albuquerque, I., Cunha, M., Lima, M.P., Galhardo, A., Maratos, F., & Gilbert, P. (2021). Building Compassionate Schools: Pilot study of a Compassionate Mind Training intervention to promote teachers' well-being. Mindfulness. https://doi.org/10.1007/s12671-021-01778-3
- [Background] Maratos, F.*, Matos, M.*, Albuquerque, I., Wood, W., Palmeira, L., Cunha, M., Lima, M.P., & Gilbert, P. (2020). Exploring the international utility of progressing Compassionate Mind Training in School Settings: A comparison of Implementation Effectiveness of the same curricula in the UK and Portugal. Psychology of Education Review, 44(2), 73-82